CLINICAL TRIAL: NCT03147300
Title: Implementation of a Best Practice Primary Health Care Model for Low Back Pain in Sweden (BetterBack): A Cluster Randomised Trial
Brief Title: Implementation of a Best Practice Primary Health Care Model for Low Back Pain
Acronym: BetterBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Allan Abbott, Associate Professor, Linkoeping University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: BetterBack
Record Dates: First submitted 2017-05-03; First posted 2017-05-10 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: Low back pain; Model of care; Primary health care; Implementation; Patient-rated outcome; Clinician-rated outcome; Cost-effectiveness
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: A cluster randomised trial with dog leg design
Who Masked: Participant
Masking Description: Participants are blinded to assignment to the control or intervention grouping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Östergötland region - Control group (Active Comparator)
  Interventions: Behavioral: Current routine practice
- Östergötland region - Intervention group (Experimental)
  Interventions: Behavioral: Multifaceted implementation of the BetterBack

INTERVENTIONS:
Behavioral: Current routine practice — Current routine practice for the primary care management of LBP
  Arms: Östergötland region - Control group
Behavioral: Multifaceted implementation of the BetterBack — The multifaceted intervention is composed of the following:
  1. Forming an implementation forum including head of departments/managers of the rehabilitation units and the clinical researchers.
  2. Forming a support team comprised of experience clinicians as local supervisors and faculty researchers as knowledge facilitators.
  3. Developing the Betterback model of care through a collaboration of the implementation forum, support team and international experts.
  4. Forming and delivering a 2-day package of education and training that the support team can utilize to assist the use of the BetterBack model of care by clinicians.
  Arms: Östergötland region - Intervention group

SUMMARY:
POPULATION: Low back pain (LBP) is a major health problem commonly requiring health care. In Sweden, primary care professionals require an evidenced based model of care for LBP.

INTERVENTION: The multi-faceted implementation of a best practice BetterBack model of care for LBP.

CONTROL: Current routine practice for LBP care before implementation of the BetterBack model of care.

OUTCOME: Patient reported measures (function, activity, health), therapist reported measures (diagnosis, intervention, specialist referral, best practice self-confidence, determinants of implementation) and cost-effectiveness.

AIM: To deliver best practice recommendations for LBP and study their most effective implementation through the BetterBack model of care.

METHOD: A cluster randomised trial with dog leg design. The hypothesis is that the BetterBack model of care will result in significantly better patient and therapist outcomes as well as cost-effectiveness compared to current routine care.

DETAILED DESCRIPTION:
Low back pain (LBP) is a major health and socioeconomic burden. LBP is usually a result of benign dysfunction and context that affects the patient's perception of pain and limits their activity and participation. At present there are no national clinical guidelines or best practice models of care in Sweden focused on the primary care of low back pain. Implementation of a model of LBP primary care based on international evidence-based guidelines is needed to improve care and patient outcomes in Sweden. This project aims to investigate the effectiveness of a best practice model of care (BetterBack) for the primary care management of LBP. A cluster randomised trial with dog leg design will be conducted in the Östergötland Health care region. The hypothesis is that the BetterBack model of care will result in significantly better patient and therapist reported outcomes as well as cost-effectiveness compared to current routine care. This by improved patient outcomes in terms of physical function, low back pain intensity, activity level, work and quality of life. Furthermore, improved care processes and knowledge support for physiotherapists can lead to a smaller proportion of patients requiring specialist care.

ELIGIBILITY:
Health care practictioner sample

Inclusion Criteria:

* Registered physiotherapists practicing in the allocated clinics and regularly working with patients with LBP

Patient sample

Inclusion Criteria:

* Males and females 18-65 years; Fluent in Swedish; Accessing public primary care due to a current episode of a first-time or recurrent debut of benign low back pain with or without radiculopathy

Exclusion Criteria:

* Current diagnosis of malignancy, spinal fracture, infection, cauda equine syndrome, ankylosing spondylitis or systemic rheumatic disease, previous malignancy during the past 5 years; Current pregnancy or previous pregnancy up to 3 months before consideration of inclusion; Patients that fulfill criteria for multimodal/multi-professional rehabilitation for complex longstanding pain; Severe psychiatric diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) for lower back related pain intensity during the latest week | Change between baseline and 3 months post baseline
  Patient rated 11-point scale consisting of integers from 0 through 10; 0 representing ''No pain'' and 10 representing ''Worst imaginable pain''
Oswestry disability index (ODI) version 2.1 | Change between baseline and 3 months post baseline
  Patient rating of LBP disability analysed as a 0 to100 scale variable where lower scores represent lower levels of low back pain disability.
Practitioner Confidence Scale (PCS) | Change between baseline and 3 months post baseline
  A total of 4 items are reported by the practitioner and a total score is collated where 4 represents greatest self-confidence and 20 represents lowest self-confidence
Incidence of participating patients recieving specialist care | 12 months after baseline
  Data on the number of participants accessing specialist care for LBP will be extracted from the Östergötland public health care region registry.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) for lower back related pain intensity during the latest week | Baseline, 3, 6 and 12 months
  Patient rated 11-point scale consisting of integers from 0 through 10; 0 representing ''No pain'' and 10 representing ''Worst imaginable pain''
Oswestry disability index (ODI) version 2.1 | Baseline, 3, 6 and 12 months
  Patient rating of LBP disability analysed as a 0 to100 scale variable where lower scores represent lower levels of low back pain disability.
The European Quality of Life Questionnaire (EQ-5D) | Baseline, 3, 6 and 12 months
  Patient rating of health-related quality of life and is computed into a 0 to 1.00 scale from worst to best possible health state by using UK index tariffs.
The Brief Illness Perception Questionnaire (BIPQ) | Baseline, 3, 6 and 12 months
  Patient rating of cognitive illness representations (consequences, outcome expectancy, personal control, treatment control, and knowledge), emotional representations (concern and emotions) as well as illness comprehensibility. An overall score 0-80 represents the degree to which the LBP is perceived as threatening or benign where a higher score reflects a more threatening view of the illness
Patient Enablement Index (PEI) | 3, 6 and 12 months
  Patient rating of enablement with a score range between 0 and 12 with a higher score intended to reflect higher patient self-care enablement
Patient satisfaction | 3, 6 and 12 months
  Patient rating of satisfaction asking "Over the course of treatment for this episode of low back pain or leg pain, how satisfied were you with the care provided by your health-care provider?" Were you very satisfied (1), somewhat satisfied (2), neither satisfied nor dissatisfied (3), somewhat dissatisfied (4), or very dissatisfied (5)?''
Patient global rating of change (PGIC) | 3, 6 and 12 months
  Patient rating of the degree of change in LBP related problems from the beginning of treatment to the present. This is measured with a balanced 11 point numerical scale.
Practitioner Confidence Scale (PCS) | Baseline, directly after commencement of implementation strategy and at 3 and 12 months afterwards
  A total of 4 items are reported by the practitioner and a total score is collated where 4 represents greatest self-confidence and 20 represents lowest self-confidence
Clinician rated health care process measures | Baseline and final clinical contact (Up to 3 months where the time point is variable depending upon the amount of clinical contact required for each patient)
  Grade of patient functional impairment and activity limitation according to the ICF brief core set for LBP is assesses by the physiotherapist where light, moderate, severe and very severe impairment/limitation is coded 0-4 respectively. A total score for baseline and an additional total score for follow-up measures at the final clinical contact (up to 3 months after baseline) is calculated from the sum of the functional impairments divided by the number of functional impairments and a similar total score is calculated for activity limitations. At the final clinical contact the therapists also report the ICD-10 diagnosis codes as well as type and number of patient treatment interventions.
Pain Attitudes and Beliefs Scale for physical therapists (PABS-PT) | Baseline, directly after education and at 3 and 12 months afterwards
  The PABS-PT consists of two factors where higher scores represent more treatment orientation regarding that factor, one measuring the biomedical treatment orientation (Score 0-60) and one regarding the biopsychosocial treatment orientation (Score 0-54)

OTHER OUTCOMES:
Determinants of implementation behavour questionnaire (DIBQ) | directly after commencement of implementation strategies and at 3 and 12 months after
  Clinician reported determinants of BetterBack implementation designed according to the Theoretical Domains Framework

CONTACTS AND LOCATIONS:
Overall Officials: Allan Abbott, Msc Physio, PhD, Principal Investigator — Linkoeping University; Birgitta Abbott, MSc Physio, PhD, Principal Investigator — Linkoeping University; Paul Enthoven, MSc Physio, PhD, Study Chair — Linkoeping University; Karin Schröder, MSc Physio, Study Chair — Linkoeping University
Locations (1):
- Östergötland health care region, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroder K, Oberg B, Enthoven P, Kongsted A, Abbott A. Confidence, attitudes, beliefs and determinants of implementation behaviours among physiotherapists towards clinical management of low back pain before and after implementation of the BetterBack model of care. BMC Health Serv Res. 2020 May 19;20(1):443. doi: 10.1186/s12913-020-05197-3. PMID 32430047
- [Derived] Abbott A, Schroder K, Enthoven P, Nilsen P, Oberg B. Effectiveness of implementing a best practice primary healthcare model for low back pain (BetterBack) compared with current routine care in the Swedish context: an internal pilot study informed protocol for an effectiveness-implementation hybrid type 2 trial. BMJ Open. 2018 Apr 24;8(4):e019906. doi: 10.1136/bmjopen-2017-019906. PMID 29691246

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03147300/Prot_SAP_000.pdf